CLINICAL TRIAL: NCT01751971
Title: Estimating Apnea Phenotypes From Routine Polysomnography: Application to Oxygen Therapy
Brief Title: Estimating Apnea Phenotypes From Polysomnography: Oxygen
Acronym: PSGtraits-O2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); American Heart Association (Other)
Responsible Party: Principal Investigator, Scott Aaron Sands, Instructor in Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2005P001296-O2PSG; R01HL090897 (NIH)
Record Dates: First submitted 2012-12-12; First posted 2012-12-18 (Estimated); Results first posted 2018-01-08 (Actual); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: Sleep Apnea
MeSH Terms: conditions — Sleep Apnea Syndromes | interventions — salicylhydroxamic acid; Air

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants were not informed whether they were breathing supplemental inspired oxygen or sham (air) on the study night. Technicians and investigators performing the study were not masked in order to carefully ensure delivery of treatment.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Inspired Oxygen First (Active Comparator): Participants breathe air with additional inspired oxygen (40%) for 1 night during an overnight sleep study (15 L/min via venturi mask). 1 week later participants will crossover to Sham (sham comparator).
  Interventions: Drug: Inspired oxygen (40%); Other: Sham
- Sham First (Sham Comparator): Participants breathe air without additional inspired oxygen for 1 night during sleep (15 L/min via Venturi mask). 1 week later participants will crossover to Inspire Oxygen (active intervention).
  Interventions: Drug: Inspired oxygen (40%); Other: Sham

INTERVENTIONS:
Drug: Inspired oxygen (40%) — Supplemental oxygen at 40% inspired via venturi mask (15 L/min). Equivalent to 5 L/min via nasal cannula.
  Other Names: Supplemental oxygen
Other: Sham — Medical air with 21% oxygen via venturi mask (15 L/min).
  Other Names: Medical air

SUMMARY:
This study seeks to employ advanced methods to estimate the individual factors contributing to sleep apnea from standard recordings made during routine clinical sleep studies. This study focuses on breathing control or "loop gain" as one of the factors contributing to sleep apnea. Increased levels of oxygen in the air is known to make breathing more stable by lowering "loop gain". Here, our goal is to use a new method capable of detecting a reduction in loop gain with oxygen. The investigators also aim to test whether a high loop gain measured at baseline/placebo predicts a greater improvement in sleep apnea with oxygen therapy.

DETAILED DESCRIPTION:
In a single-blinded randomized crossover study, inspired oxygen/air (40%/21%) is delivered on two separate nights. Loop gain is measured from routine polysomnography using a novel mathematical method. A value of loop gain >1 reflects unstable breathing, and a value less than but approaching 1 denotes a system more prone to oscillate. Loop gain is measured as the changes in ventilatory drive/effort that arises subsequent to changes in ventilation (e.g. due to obstructive apnea). A simple chemoreflex model (gain, time constant, delay) is fit to surrogate ventilation data (derived from airflow) during sleep. The best model is one that best matches the elevated ventilatory drive (measured as ventilation in the absence of airflow obstruction) based on the prior apneic/hypopneic fall in ventilation. Loop gain is calculated from this model. We aim to use loop gain measured on and off oxygen to determine whether a strong response (reduction in apnea severity) can be predicted by a higher loop gain (in the sham arm) using our method. We also assessed whether assessing upper airway anatomy/collapsibility, dilator muscle responsiveness, and the arousal threshold helped to predict responses to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Apnea/hypopnea index >20 events per hour
* Age 20-79 years

Exclusion Criteria:

* COPD with desaturation (resting SpO2<96%)
* Use of respiratory stimulants or depressants
* Pregnancy

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2012-11; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: SCOTT A Sands, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Sands SA, Edwards BA, Terrill PI, Butler JP, Owens RL, Taranto-Montemurro L, Azarbarzin A, Marques M, Hess LB, Smales ET, de Melo CM, White DP, Malhotra A, Wellman A. Identifying obstructive sleep apnoea patients responsive to supplemental oxygen therapy. Eur Respir J. 2018 Sep 27;52(3):1800674. doi: 10.1183/13993003.00674-2018. Print 2018 Sep. PMID 30139771

RESULTS

PARTICIPANT FLOW:
Groups:
- Oxygen First: Participants participate in inspired oxygen arm (40% oxygen) first, then the air night (21% oxygen) second
  Inspired oxygen (40%): Supplemental oxygen at approximately 40% e.g. via Pink venturi mask
- Air First: Participants participate in the air night (sham) first, then the oxygen night second.
  Sham: Medical air with 21% oxygen e.g. via Pink venturi mask
Period: Overall Study
Arm/Group | Oxygen First | Air First
Started | 22 | 25
Completed | 20 | 24
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oxygen First | Air First | Total
Number analyzed (Participants) | 22 | 25 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (13) | 49 (22) | 52 (19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 10 | 15
  Male | 17 | 15 | 32

OUTCOME MEASURES:

1. Primary Outcome: Apnea-hypopnea Index
Description: Apnea-hypopnea index (AHI) will be compared between oxygen and sham nights. Hypopneas are based on 30% reduction in airflow (no desaturation or arousal criteria). AHI data are exclusive to non-REM supine sleep.
  The results presented here are for the AHI at each intervention ("per intervention") regardless of the sequence (preferred clinicaltrials.gov format).
  Please note, however, that the a priori outcome measure was the reduction in AHI with oxygen as a percent of sham values, i.e. (AHI on sham - AHI on oxygen)/(AHI on sham) % (a comparison with greater statistical power), compared between patient subgroups (see Statistical Analysis section).
  Subgroups were defined a priori as higher (>=0.7) versus lower loop gain (<0.7), but tests were also performed in subgroups defined by "favorable" versus "unfavorable" pathophysiology.
Time Frame: 1 night
Population: Patients with AHI>20
Measure: Mean (Standard Error); unit: events/hour
Groups:
- Inspired Oxygen: Inspired oxygen (40%) for 1 night via venturi mask.
- Sham: Sham: Medical air with 21% oxygen via venturi mask
Arm/Group | Inspired Oxygen | Sham
Number analyzed (Participants) | 36 | 36
events/hour
  All patients | 40.5 (3.8) | 57.9 (3.7)
  Patients with high loop gain (LG1): number analyzed (Participants) | 13 | 13
  Patients with high loop gain (LG1) | 48.5 (6.4) | 74.3 (6.1)
  Patients with low loop gain (LG1): number analyzed (Participants) | 23 | 23
  Patients with low loop gain (LG1) | 35.9 (4.6) | 48.5 (3.4)
  Patients with favorable pathophysiology: number analyzed (Participants) | 14 | 14
  Patients with favorable pathophysiology | 22.5 (4.3) | 49.5 (4.8)
  Patients with unfavorable pathophysiology: number analyzed (Participants) | 21 | 21
  Patients with unfavorable pathophysiology | 51.9 (4.1) | 63.2 (5.0)
Statistical Analysis 1: Comparison: Inspired Oxygen vs Sham; Primary statistical comparison was the percent reduction in AHI----[AHI(sham)-AHI(oxygen)]/AHI(sham) %----between two phenotypic patient subgroups. Patient subgroups were defined by the loop gain (LG1) measured on the sham night as "high" or "low" (a priori cutoff LG1=0.7); Test type: Superiority; p = 0.4, t-test, 2 sided; Mean Difference (Net) = 10.5, 95% CI 2-sided [-16 to 37.1] — Positive estimated value would represent a greater reduction in AHI with oxygen (% sham) in the high vs low loop gain group
Statistical Analysis 2: Comparison: Inspired Oxygen vs Sham; Here we aimed to confirm that there was a difference between AHI on oxygen vs sham (overall, i.e. in unselected patients). This test, however was not part of our primary objective; Test type: Superiority; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = 17.4, 95% CI 2-sided [10.7 to 24.1], Standard Error of Mean 3.3 — Direction of comparison: Positive estimation parameter would indicate lower AHI on oxygen versus sham
Statistical Analysis 3: Comparison: Inspired Oxygen vs Sham; The primary goal of the study was to identify a phenotypic subgroup of patients with sleep apnea that responds preferentially to oxygen (percent reduction in AHI----[AHI(sham)-AHI(oxygen)]/AHI(sham) %). We defined patient subgroups ("favorable" versus "unfavorable") based on the four key phenotypic traits (loop gain, collapsibility, arousal threshold, muscle responses) measured on the sham night, with the use of multiple logistic regression and leave-one-out cross validation; Test type: Superiority; p = 0.001, t-test, 2 sided; Mean Difference (Net) = 42.8, 95% CI 2-sided [21.0 to 64.6] — Direction of comparison: Positive estimated value would indicate a greater percentage reduction in AHI (oxygen vs. sham) in favorable vs. unfavorable subgroups

2. Secondary Outcome: Frequency of EEG Arousals (Events Per Hour)
Description: Frequency of scored EEG arousals per hour of non-REM sleep. Note: Our objective was to describe changes in secondary outcomes within phenotypic subgroups. Overall effects (unselected patients / ignoring phenotypic subgroups) are first presented below, followed by effects in favorable vs. unfavorable subgroups.
Time Frame: 1 night
Population: Patients with AHI>20
Measure: Mean (Standard Error); unit: events/hr
Groups:
- Inspired Oxygen: Inspired oxygen (40%): Supplemental oxygen at approximately 40% e.g. via Pink venturi mask
- Sham: Sham: Medical air with 21% oxygen e.g. via Pink venturi mask
Arm/Group | Inspired Oxygen | Sham
Number analyzed (Participants) | 36 | 36
events/hr
  All patients | 35.9 (3.4) | 50.3 (3.7)
  Patients with favorable pathophysiology: number analyzed (Participants) | 14 | 14
  Patients with favorable pathophysiology | 20.8 (3.0) | 39.7 (5.1)
  Patients with unfavorable pathophysiology: number analyzed (Participants) | 22 | 22
  Patients with unfavorable pathophysiology | 45.4 (4.1) | 57.0 (4.6)

3. Secondary Outcome: Overnight Change in Systolic Blood Pressure
Description: The change in systolic blood pressure overnight. Two supine oscillometric measurements of blood pressure are made: just prior to lights out (evening), and after lights on (morning).
Time Frame: 1 night
Population: Patients with AHI>20
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Inspired Oxygen | Sham
Number analyzed (Participants) | 36 | 36
mmHg
  All patients | -0.8 (1.4) | 3.0 (1.9)
  Patients with favorable pathophysiology: number analyzed (Participants) | 14 | 14
  Patients with favorable pathophysiology | -2.8 (1.9) | 3.4 (2.9)
  Patients with unfavorable pathophysiology: number analyzed (Participants) | 22 | 22
  Patients with unfavorable pathophysiology | 0.5 (1.9) | 2.8 (2.5)

4. Secondary Outcome: Overnight Change in Diastolic Blood Pressure
Description: The change in diastolic blood pressure overnight. Two supine oscillometric measurements of blood pressure are made: just prior to lights out (evening), and after lights on (morning).
Time Frame: 1 night
Population: Patients with AHI>20
Measure: Mean (Standard Error); unit: mmHg
Groups:
- Inspired Oxygen: Inspired oxygen (40%) for 1 night via venturi mask. "Arm" here is defined as the Oxygen Intervention. 18 participants participated in inspired oxygen arm (40% oxygen) first, then the air night (21% oxygen) second. 18 participants participated in the other order.
- Sham: Sham: Medical air with 21% oxygen e.g. via Pink venturi mask "Arm" here is defined as the Sham Intervention. 18 participants participated in inspired oxygen arm (40% oxygen) first, then the air night (21% oxygen) second. 18 participants participated in the other order.
Arm/Group | Inspired Oxygen | Sham
Number analyzed (Participants) | 36 | 36
mmHg
  All patients | 0.9 (0.9) | 4.1 (1.5)
  Patients with favorable pathophysiology: number analyzed (Participants) | 14 | 14
  Patients with favorable pathophysiology | -0.7 (1.2) | 6.4 (2.3)
  Patients with unfavorable pathophysiology: number analyzed (Participants) | 22 | 22
  Patients with unfavorable pathophysiology | 2.0 (1.2) | 2.5 (2.0)

5. Secondary Outcome: Subjective Sleep Quality (Oxygen vs Sham)
Description: Better(+1)/Same(0)/Worse(-1) on oxygen vs sham, i.e. "a relative comparison between arms". When subjects had completed the entire study, they were asked to compare subjectively their sleep quality on the first versus second study.
Time Frame: 1 night
Population: Patients with AHI>20. One patient, whose treatment and sham nights were separated by an extended duration (due to scheduling), did not provide data for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- All Participants: Data are presented as a single arm because results are inherently a comparison between arms. Participants were asked to rate whether their sleep quality was better/same/worse on study night 2 versus study night 1. Data are presented in terms of better/same/worse on oxygen compared to sham.
Arm/Group | All Participants
Number analyzed (Participants) | 35
units on a scale
  All patients | 0.34 (0.13)
  Patients with favorable pathophysiology: number analyzed (Participants) | 13
  Patients with favorable pathophysiology | 0.69 (0.17)
  Patients with unfavorable pathophysiology: number analyzed (Participants) | 22
  Patients with unfavorable pathophysiology | 0.14 (0.18)

6. Secondary Outcome: Subjective Sleepiness/Alertness (Stanford Sleepiness Scale)
Description: Assessed in the morning after the single night of treatment. Minimum score: 1 (alert), maximum score: 7 (not alert).
Time Frame: 1 night
Population: Patients with AHI>20
Measure: Mean (Standard Error); unit: Scores on a scale
Groups:
- Inspired Oxygen: Inspired oxygen (40%) via Pink venturi mask
Arm/Group | Inspired Oxygen | Sham
Number analyzed (Participants) | 36 | 36
Scores on a scale
  All patients | 2.13 (0.19) | 2.03 (0.18)
  Patients with favorable pathophysiology: number analyzed (Participants) | 14 | 14
  Patients with favorable pathophysiology | 2.14 (0.32) | 2.11 (0.26)
  Patients with unfavorable pathophysiology: number analyzed (Participants) | 22 | 22
  Patients with unfavorable pathophysiology | 2.13 (0.25) | 1.99 (0.25)

ADVERSE EVENTS:
Groups:
- Inspired Oxygen: Inspired Oxygen 40%
- Sham: Sham, room air
Arm/Group | Inspired Oxygen | Sham
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/45
Other Adverse Events (participants affected / at risk) | 0/46 | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes